CLINICAL TRIAL: NCT01003132
Title: A Pilot Randomised Controlled Trial of Acceptance and Commitment Therapy for Distress Following Psychosis
Brief Title: Assessing the Effectiveness of Acceptance and Commitment Therapy for Distress Following Psychosis
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Dr Ross White/Clinical Research Fellow, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PN09CP213; Ethics Ref:09/S0701/74
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Psychosis; Schizophrenia; Bipolar Disorder; Schizo-affective Disorder
Keywords: Psychosis; Distress; Mindfulness; Acceptance; Values
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment As Usual (No Intervention): Treatment as usual as determined by the clinical team responsible for the individual's care
- Acceptance and Commitment Therapy (Active Comparator): Up to 10 sessions of Acceptance and Commitment Therapy plus treatment as usual
  Interventions: Other: Acceptance and Commitment Therapy

INTERVENTIONS:
Other: Acceptance and Commitment Therapy — Up to 10 sessions of a psychological therapy called Acceptance and Commitment Therapy
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy

SUMMARY:
This research investigates a new talking therapy aimed at helping people to come to terms with the experience of psychosis. The new therapy is called Acceptance and Commitment Therapy for psychosis (PACT). PACT aims to help people:

1. Develop a sense of "mindfulness." Mindfulness allows you to be fully aware of your here-and-now experience, with an attitude of openness and curiosity. It is hoped that this will help reduce the impact of painful thoughts and feelings.
2. Take effective action that is conscious and deliberate, rather than impulsive. It is hoped that this will allow people to be motivated, guided, and inspired by the things that they value in life.

It is hoped that PACT will help to reduce the level of distress that individuals diagnosed with psychosis have been experiencing and help them to stay well in the future.

DETAILED DESCRIPTION:
Emphasis has been placed on treating the 'positive symptoms' of psychosis (e.g. hallucinations and delusions). Concordance rates with anti-psychotic medication can be low. Even when positive symptoms are successfully treated, emotional distress can remain e.g. depression, anxiety and trauma. Relapse occurs in up to two thirds of patients within two years of the first episode. The treatment of subsequent episodes has been shown to be progressively less efficacious. Research has shown that fear of recurrence patients can experience following psychosis is predictive of relapse. Randomised clinical trials have found that Cognitive Behaviour Therapy (CBTp) is efficacious for treating residual distressing positive and negative symptoms. However, the evidence for treating emotional dysfunction (e.g. social anxiety, post-psychotic depression) is less clear. Acceptance and Commitment Therapy (ACT) incorporates acceptance and mindfulness elements into a CBT framework. Rather than altering the content or frequency of cognitions, ACT seeks to alter the individual's psychological relationship with thoughts, feelings and sensations to promote psychological flexibility. This research will be a pilot randomised control trial of ACT for treating distress following psychosis. This pilot study will establish (a) whether a larger scale multi-centre randomised controlled trial is warranted, (b) the acceptability of Acceptance and Commitment Therapy (c) the expected primary and secondary outcomes for such a trial and (d) the sample size required to detect such outcomes. It is hypothesised that ACT plus treatment as usual will be associated with a greater reduction in levels of distress than treatment as usual only.

ELIGIBILITY:
Inclusion Criteria:

* Participants will meet DSM-IV-TR (APA, 2000) criteria for a psychotic disorder determined by a diagnosis of a psychotic disorder (i.e., Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder, Delusional Disorder, Brief Psychotic Disorder, Psychotic Disorder NOS) or Bipolar Disorder (with psychotic features).
* Participants will also be aged 18-65

Exclusion Criteria:

* Participants will be excluded if there is a

  * diagnosis of learning disability
  * inability to participate in psychotherapy/research due to acute medical condition or florid psychosis (as defined by a score of 5 or over on the Positive Syndrome scale of the PANSS)
  * psychotic symptoms due to a general medical condition
  * they are receiving a systematic psychological therapy at the point of recruitment/randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Measuring change in depression and anxiety | Baseline and 3 month follow-up
  The Hospital Anxiety and Depression Scale
Changes in believability, distress and frequency of positive symptoms | Baseline and up to 9 months follow-up

SECONDARY OUTCOMES:
Measuring change in mindfulness skills and psychological flexibility | Baseline and up to 9 month follow-up
  The Kentucky Inventory of Mindfulness Skills, The Acceptance and Action Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ross G White, BSc, PhD, DClinPsy, Principal Investigator — University of Glasgow
Locations (1):
- Greater Glasgow and Clyde NHS, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Background] Bach P, Hayes SC. The use of acceptance and commitment therapy to prevent the rehospitalization of psychotic patients: a randomized controlled trial. J Consult Clin Psychol. 2002 Oct;70(5):1129-39. doi: 10.1037//0022-006x.70.5.1129. PMID 12362963
- [Background] Gaudiano BA, Herbert JD. Acute treatment of inpatients with psychotic symptoms using Acceptance and Commitment Therapy: pilot results. Behav Res Ther. 2006 Mar;44(3):415-37. doi: 10.1016/j.brat.2005.02.007. PMID 15893293
- [Background] Hayes, S.C., Strosahl, K. and Wilson, K.G. (1999). Acceptance and Commitment Therapy: An experiential approach to behavior change, The Guilford Press, New York